CLINICAL TRIAL: NCT00030680
Title: Phase II Pilot Study Of Moderate Dose Radiotherapy For Inoperable Aggressive Fibromatoses
Brief Title: Radiation Therapy in Treating Patients With Aggressive Fibromatoses
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-62991-22998; EORTC-62991; EORTC-22998
Record Dates: First submitted 2002-02-14; First posted 2003-01-27 (Estimated); Last update posted 2013-08-27 (Estimated); Status verified 2013-08

CONDITIONS: Desmoid Tumor
Keywords: desmoid tumor
MeSH Terms: conditions — Desmoid Tumors | interventions — Radiotherapy

INTERVENTIONS:
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells.

PURPOSE: Phase II trial to study the effectiveness of radiation therapy in treating patients who have aggressive fibromatoses.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of moderate-dose radiotherapy, in terms of local control, in patients with aggressive fibromatoses.
* Determine the acute and late side-effects of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive radiotherapy 5 days a week for 5.5 weeks for a total of 56 Gy in 28 fractions.

Patients are followed every 3 months for 2 years and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed aggressive fibromatoses arising in any site

  * Primary, recurrent, or progressive disease that is inoperable or requires a major operation resulting in a large functional or cosmetic deficit or mutilation

    * Progressive disease defined as at least 20% increase in tumor size on 2 MRI scans within 1 year after any prior therapy except radiotherapy OR
  * Incompletely resected tumor with gross residual disease not suitable for further surgery

    * Resected within the past 3 months
* Lesions must be suitable for radiotherapy

  * No bulky intra-abdominal disease in close relation to small bowel
* Measurable disease

PATIENT CHARACTERISTICS:

Age:

* 16 and over

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No conditions that would preclude study follow-up

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Prior chemotherapy allowed
* No concurrent chemotherapy

Endocrine therapy:

* Prior endocrine therapy allowed
* No concurrent endocrine therapy

Radiotherapy:

* See Disease Characteristics
* No prior radiotherapy to indicator lesion

Surgery:

* See Disease Characteristics
* Prior surgery allowed

Other:

* No prior isolated limb perfusion with tumor necrosis factor
* No concurrent isolated limb perfusion with tumor necrosis factor

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2001-11; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Local control as assessed by MRI at 3 years

SECONDARY OUTCOMES:
Toxicity as assessed by CTC 2.0
Response as assessed by MRI

CONTACTS AND LOCATIONS:
Overall Officials: R. B. Keus, MD, Study Chair — Arnhems Radiotherapeutisch Instituut; Thomas Schnabel, MD, Study Chair — Klinikum der Stadt Ludwigshafen am Rhein
Locations (21):
- Belgium (2):
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
- France (3):
  - Institut Bergonie, Bordeaux
  - Centre Leon Berard, Lyon
  - CHU de la Timone, Marseille
- Southwest German Cancer Center at Eberhard-Karls-University, Tübingen, Germany
- Netherlands (6):
  - Arnhems Radiotherapeutisch Instituut, Arnhem
  - University Medical Center Groningen, Groningen
  - Leiden University Medical Center, Leiden
  - Maastro Clinic - Locatie Maastricht, Maastricht
  - Daniel Den Hoed Cancer Center at Erasmus Medical Center, Rotterdam
  - Dr. Bernard Verbeeten Instituut, Tilburg
- Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Warsaw, Poland
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland
- United Kingdom (7):
  - Queen Elizabeth Hospital at University Hospital of Birmingham NHS Trust, Birmingham, England
  - Cookridge Hospital, Leeds, England
  - Christie Hospital, Manchester, England
  - Mount Vernon Cancer Centre at Mount Vernon Hospital, Northwood, England
  - Nottingham City Hospital NHS Trust, Nottingham, England
  - Cancer Research Centre at Weston Park Hospital, Sheffield, England
  - Royal Marsden - Surrey, Sutton, England